CLINICAL TRIAL: NCT01151722
Title: Adjuvant Intravitreal Bevacizumab in Pars Plana Vitrectomy for Diabetic Vitreous Hemorrhage
Acronym: ABeVi
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: USP, USP
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HCRP22
Record Dates: First submitted 2010-06-25; First posted 2010-06-28 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-02

CONDITIONS: Recurrent; Hemorrhage
MeSH Terms: conditions — Recurrence; Hemorrhage | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- no injection (No Intervention): no bevacizumab
- experimental 2 (Experimental): bevacizumab before vitrectomy
  Interventions: Procedure: bevacizumab injection
- experimental 3 (Experimental): bevacizumab after vitrectomy
  Interventions: Procedure: bevacizumab injection

INTERVENTIONS:
Procedure: bevacizumab injection — bevacizumab injection before vitrectomy
  Arms: experimental 2
Procedure: bevacizumab injection — bevacizumab injection after vitrectomy
  Arms: experimental 3

SUMMARY:
Postoperative vitreous hemorrhage is a common complication after vitrectomy for proliferative diabetic retinopathy. There have been efforts to lower the incidence of postoperative vitreous hemorrhage such as preoperative bevacizumab injection. Bevacizumab (Avastin) is a potent inhibitor of angiogenesis and has been shown to decrease retinal and iris neovascularization in proliferative diabetic retinopathy. Recently there have been reports showing that preoperative bevacizumab injection could reduce intraoperative bleeding from abnormal vessels and could make surgery easier and more successful. Our hypothesis is that intraoperative bevacizumab injection could reduce postoperative vitreous hemorrhage by inhibiting the vessel formation after surgery.

We started the prospective randomized comparative study to determine the effect of pre and intra-operative bevacizumab injection on postoperative vitreous hemorrhage after diabetic vitrectomy in comparison to vitrectomy without any adjuvant drug.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing first vitrectomy for vitreous hemorrhage secondary to proliferative diabetic retinopathy

Exclusion Criteria:

* follow-up period of less than 3 months
* not first vitrectomy
* abnormal blood coagulation
* uncontrolled hypertension

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Vitreous hemorrhage recurrence | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas de Ribeirão Preto - University of São Paulo, Ribeirão Preto, São Paulo, Brazil

REFERENCES:
- [Derived] Dervenis P, Dervenis N, Smith JM, Steel DH. Anti-vascular endothelial growth factors in combination with vitrectomy for complications of proliferative diabetic retinopathy. Cochrane Database Syst Rev. 2023 May 31;5(5):CD008214. doi: 10.1002/14651858.CD008214.pub4. PMID 37260074